CLINICAL TRIAL: NCT01841879
Title: Mumbai Worksite Tobacco Control Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Healis-Sekhsaria Institute for Public Health (Other); Carelon Research (Other); Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Glorian Sorensen, Professor of Society, Human Development, and Health, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01CA140304 (NIH); R01CA140304 (NIH)
Record Dates: First submitted 2013-03-19; First posted 2013-04-29 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2017-04

CONDITIONS: Tobacco Use Cessation
MeSH Terms: conditions — Tobacco Use Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Program (Experimental): Receives the full Healthy, Safe, and Tobacco-Free Worksites intervention
  Interventions: Behavioral: Intervention Program
- Delayed Intervention Control (Other): Receives abbreviated 2-month delayed intervention designed to provide employees with knowledge and skills to quit tobacco after final data collection time point, as well as one non-tobacco event in between data collection points.
  Interventions: Behavioral: Delayed Intervention

INTERVENTIONS:
Behavioral: Intervention Program — Receives an integrated tobacco control and occupational health (OH) intervention (The Healthy, Safe, and Tobacco-Free Worksites program) aimed at promoting tobacco cessation among workers and supporting the adoption, implementation, and enforcement of tobacco control policies.
  Through six health education events at the worksites, blue-collar workers (who face dual health risks through their exposures to occupational hazards and their high rates of tobacco use) will gain the knowledge, skills, and social support needed to quit tobacco use.
  Simultaneously, management will receive OH and tobacco policy consultations to help build a healthy and safe work environment, where workers' hazardous exposures are reduced.
  Other Names: Healthy, Safe, and Tobacco-Free Worksites Program
  Arms: Intervention Program
Behavioral: Delayed Intervention — Receives abbreviated 2-month delayed intervention designed to provide employees with knowledge and skills to quit tobacco after final data collection time point, as well as one non-tobacco event in between data collection points.
  Arms: Delayed Intervention Control

SUMMARY:
The investigators are designing and testing the effectiveness of an integrated tobacco control and occupational health (OH) intervention aimed at promoting tobacco cessation among workers and supporting the adoption, implementation, and enforcement of tobacco control policies in 20 manufacturing worksites in the greater Mumbai region of India.

DETAILED DESCRIPTION:
Through 6 health education events at the worksites, blue-collar workers (who face dual health risks through their exposures to occupational hazards and their high rates of tobacco use) will gain the knowledge, skills, and social support needed to quit tobacco use.

Simultaneously, management will receive OH and tobacco policy consultations to help build a healthy and safe work environment, where workers' hazardous exposures are reduced.

ELIGIBILITY:
Inclusion Criteria:

* Manufacturing worksites located in the Mumbai, Thane, or Raigad districts of India
* Employ at least 60% production workers/40% administrative staff OR at employ at least 200 production workers on staff. NOTE: We are defining "workers" as anyone who is on the company roster, regardless of whether they're permanent or contractual
* Companies must be autonomous decision-makers and allow us to function at their worksite
* Companies must be willing to provide us with a current employee roster

Exclusion Criteria:

* Employees do not speak English, Hindi, or Marathi

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 6880 (Actual)
Dates: Start 2010-06; Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
Tobacco use cessation | 6-month post intervention

SECONDARY OUTCOMES:
Changes in company tobacco policy | 6-month post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Glorian Sorensen, PhD, MPH, Principal Investigator — Harvard School of Public Health, Dana-Farber Cancer Institute
Locations (1):
- Healis-Sekhsaria Institute for Public Health, Navi Mumbai, Maharshtra, India

REFERENCES:
- [Derived] Sorensen G, Pednekar M, Cordeira LS, Pawar P, Nagler EM, Stoddard AM, Kim HY, Gupta PC. Effects of a worksite tobacco control intervention in India: the Mumbai worksite tobacco control study, a cluster-randomised trial. Tob Control. 2017 Mar;26(2):210-216. doi: 10.1136/tobaccocontrol-2015-052671. Epub 2016 Feb 16. PMID 26883793
- See also: Healis-Sekhsaria Institute for Public Health's website — http://www.healis.org
- See also: The Center for Community-Based Research's website — http://www.community-based-research.org/